CLINICAL TRIAL: NCT04925492
Title: Positron Emission Tomography (PET) Imaging of Vaso-occlusive Crisis(VOC) in Sickle Cell Disease (SCD).
Brief Title: PET Imaging of Vaso-Occlusive Crisis (VOC) in SCD
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Enrico Novelli (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Enrico Novelli, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: STUDY20020135; R01HL154629 (NIH)
Record Dates: First submitted 2020-12-15; First posted 2021-06-14 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Sickle Cell Disease
Keywords: PET MRI
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Intervention Model Description: Population of adult Sickle Cell patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Finding Optimal Scan Timing (Experimental): Group A will receive two PET scans after the radiotracer injection to learn the best timing of the scan for the rest of the people in the study during participant's baseline state. Participants will receive another injection of the radiotracer during a sickle cell crisis and have one PET scan. Receive an optional injection and perform another PET scan 12 months after your sickle cell crisis if there were technical problems the previous scans.
  Interventions: Radiation: Positron Emission Tomography; Drug: Cu-64]-LLP2A
- Scan at Determined Optimal Timepoint (Experimental): Group B participants will receive an injection of the radiotracer and undergo only one PET scan during a baseline state. Participants will receive another injection of the radiotracer during a sickle cell crisis and have one PET scan. Receive an optional injection and perform another PET scan 12 months after your sickle cell crisis if there were technical problems the previous scans.
  Interventions: Radiation: Positron Emission Tomography; Drug: Cu-64]-LLP2A

INTERVENTIONS:
Radiation: Positron Emission Tomography — An imaging method that uses radiotracers to view changes in the metabolic process.
  Other Names: PET Scan
Drug: Cu-64]-LLP2A — A radioactive tracer used in PET imaging.
  Other Names: Cu-64]-LLP2A Radiotracer

SUMMARY:
The purpose of this study is to find objective biomarkers of vaso-occlusion (blood vessel blockage) in people with SCD. Using information from earlier studies and work being done, researchers have developed a strategy to image VOC, using positron emission tomography (PET).

The ability to see and measure VOC in SCD patients can help patient care, by showing when and how a VOC is occurring or going to occur. Studying this method will also help in future drug research, as it will allow researchers to deliver promising new medications that target hyper-adhesion and sickling in people with SCD.

DETAILED DESCRIPTION:
The purpose of this study is to find objective biomarkers of vaso-occlusion (blood vessel blockage) in people with Sickle Cell Disease(SCD). Using information from earlier studies, and work being done at Washington University, a strategy to image vaso-occulusive crisis (VOC) has been developed, using positron emission tomography (PET) for anatomical localization only. 64Cu-LLP2A is the radio tracer used for the study.

Aim: To develop quantitative PET imaging of VOC in patients with SCD. The researchers hypothesize that the radio tracer 64Cu-LLP2A uptake increases proportionally to the intensity of pain in patients with VOC, compared to baseline values. This increase in uptake will be assessed focally in areas of pain as well as globally to reflect heightened systemic inflammation.

Primary and secondary study endpoint: The overarching hypothesis of this study is that PET tracer uptake of intensity of 64Cu-LLP2A is a real time, quantitative measure of hyper adhesion in VOC.

ELIGIBILITY:
Inclusion Criteria:

* Have a confirmed diagnosis of SCD (HbSS, SC, S/β-thalassemia, SD, SE, SO) by hemoglobin electrophoresis/High Performance Liquid Chromatography (HPLC)
* Aged 18 and above
* Ability to understand and provide informed consent.
* If receiving hydroxyurea or L-glutamine, crizanlizumab, voxelotor or erythropoietin stimulating agents, must have been receiving the drug for at least 12 weeks prior to screening and plan to continue taking the drug at the same dose and schedule during the study
* Experienced at least 2 VOCs leading to healthcare visit within the 12 months prior to screening visit as determined by medical history.

Exclusion Criteria:

* Active malignancy
* Current pregnancy or breast feeding
* Participating in a chronic transfusion program (pre-planned series of transfusions for prophylactic purposes) and/or planning on undergoing an exchange transfusion during the duration of the study; episodic transfusion in response to worsened anemia or VOC is permitted
* Received active treatment on another investigational trial within 30 days (or 5 half-lives of that agent, whichever is greater) prior to screening visit or plans to participate in another investigational drug trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-11-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in PET tracer uptake in VOC | Up to five years from first assessment depending on when VOC occurs.
  Intensity of PET tracer uptake in VOC will be measured and compared to uptake at baseline in predefined regions of interest and over the whole body
Association of PET tracer uptake with intensity of pain in VOC | 2 hours during an assessment while in VOC.
  Intensity of PET tracer uptake will be compared to intensity of pain by Visual Analog Score (scored from 0-10, with 0 meaning no pain, and 10 meaning the most pain) and pain characteristic assessed by the Painimation assessment tool in specific anatomical areas in the patients during a sickle cell vaso-occlusive event.
Association of PET tracer uptake with clinical VOC markers | Up to the length of a hospital visit for treatment of VOC. On average, about 5 days.
  Measure of PET tracer uptake will be compared with clinical markers of vaso-occlusive events including length of stay and hematologic markers of hemolysis.

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Novelli, MD, MS, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Information and stored samples may be shared without identifiers with other researchers in the future. These researchers will not receive identifiable information linking data or sample back to individual participants. This access may be granted for the advancement of scientific knowledge. Any future sharing will be conducted under an approved sharing agreement